CLINICAL TRIAL: NCT04772183
Title: OxyGap : Comparison Between Different Pulse Oximeter and With the Arterial Blood
Brief Title: OxyGap : Comparison Between Different Pulse Oximeter and With the Arterial Blood Gase
Acronym: OxyGap
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal investigator, Laval University
Other Study IDs: 2021-3624
Record Dates: First submitted 2021-02-17; First posted 2021-02-26 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Failure; Hypoxemia; Hyperoxemia
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: SpO2 and SaO2 comparison — Several pulse oximeter will be place on patient find few minutes before arterial blood gases.
  During an arterial blood sample, all SpO2 will be recorded

SUMMARY:
The oximeter is used to monitor intensive care patients undergoing oxygen therapy. It indicates pulsed oxygen saturation (SpO2), a reflection of arterial oxygen saturation (SaO2) which enables detection of hypoxemia and hyperoxia, both deleterious state. Current SpO2 recommendations aim to reduce both risk of hypoxemia and hyperoxia. SpO2 is considered the 5th vital sign.

Current recommendations for SpO2 targets do not consider the variability of oximeters used in clinical practice. This variability and lack of specification represent an obstacle to an optimal practice of oxygen therapy.

Thus, this study aims to compare the SpO2 values of different oximeters (Nonin, Masimo, Philips, Nellcor) used in clinical practice with the SaO2 reference value obtained by an arterial gas in order to specify the precision and the systematic biases of the oximeters studied. This data will also make it possible to refine the recommendations concerning optimal oxygenation

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Patients admitted to the Intensive Care Unit
* Artery catheter already installed

Exclusion Criteria:

* No signal with the oximeter
* Pigmented nails or nail polish
* Methemoglobinemia
* Patient in isolation (multi-resistant bacteria, C-Difficile, COVID-19…)
* Prone position

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patient in ICU with arterial catheter already installed will be consider.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Diffence between Nellcor SpO2 and the SaO2 value | During arterial blood gase sample
  Diffence between Nellcor oximeter SpO2 and the SaO2 value
Diffence between FreeO2 SpO2 and the SaO2 value | During arterial blood gase sample
  Diffence between Nonin (FreeO2) oximeter SpO2 and the SaO2 value
Diffence between Nonin ear clip and the SaO2 value | During arterial blood gase sample
  Diffence between Nonin (ear sensor) oximeter SpO2 and the SaO2 value
Diffence between Masimo SpO2 and the SaO2 value | During arterial blood gase sample
  Diffence between Masimo oximeter SpO2 and the SaO2 value
Diffence between Philips SpO2 and the SaO2 value | During arterial blood gase sample
  Diffence between Philips oximeter SpO2 and the SaO2 value
Diffence between Contec SpO2 and the SaO2 value | During arterial blood gase sample
  Difffence between Contec oximeter SpO2 and the SaO2 value
Diffence between Bejing choice SpO2 and the SaO2 value | During arterial blood gase sample
  Diffence between Bejing choice oximeter SpO2 and the SaO2 value

SECONDARY OUTCOMES:
Overestimation and underestimation of SaO2 | During arterial blood gase sample
  % of pairs with overestimation and underestimation of SaO2 for each oximeter.
Hypoxemia detection | During arterial blood gase sample
  Ability to detect hypoxemia (SpO2 below 90% and PaO2 < 60 mmHg)
Hyperoxemia detection | During arterial blood gase sample
  Ability to detect hyperoxemia (SpO2 above 95% and PaO2 > 100 mmHg)
Gaps between the different oximeters | During arterial blood gase sample
  Average of the SpO2 value gaps between the different oximeters tested
Finger and ear sensor comparison | During arterial blood gase sample
  Comparison of the finger sensor and ear clip sensor for Nonin oximeter

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CHUM, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec

IPD SHARING:
Plan to Share IPD: No